CLINICAL TRIAL: NCT03411382
Title: Influence of Sit Muscle Strength Training and Game on Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Taiwan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Chiu Shu-Ching, Principal investigator of nursing department, Central Taiwan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CentralTaiwanUST
Record Dates: First submitted 2017-12-09; First posted 2018-01-26 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Aging; Physical Disability; Dementia; Elderly
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sit muscle strength training (Experimental): Sit muscle strength training using a sand bag grip ball conducted twice a week. Each exercise session will begin and end with a 5-15 minute warm-up and cool-down routine. The exercise program consists of 20-40 minute chair-based resistance exercises.
  Interventions: Other: Sit muscle strength training
- Game training (Experimental): Game training (including ball activities, clay courses, massage, puzzles, painting conducted four times a week). Each section 30-60 minutes.
  Interventions: Other: Game training
- Sitting strength + game training (Experimental): Sitting strength training (using sandbag training conducted twice a week) and game training (such as ball activities and clay courses) conducted twice a week).
  Interventions: Other: Sitting strength + game training
- Health education (Placebo Comparator): Health education (conducted once a month). Each section 50-60 minutes. The topics are oral hygiene, medicine safe, living safe, food safe.
  Interventions: Other: Health education

INTERVENTIONS:
Other: Sit muscle strength training — Sit muscle strength training using a sand bag grip ball conducted twice a week. Each exercise session will begin and end with a 5-15 minute warm-up and cool-down routine. The exercise program consists of 20-40 minute chair-based resistance exercises.
  Arms: Sit muscle strength training
Other: Game training — Game training (including ball activities, clay courses, massage, puzzles, painting conducted four times a week). Each section 30-60 minutes.
  Arms: Game training
Other: Sitting strength + game training — Sitting strength training (using sandbag training conducted twice a week) and game training (such as ball activities and clay courses) conducted twice a week).
  Arms: Sitting strength + game training
Other: Health education — Health education (conducted once a month). Each section 50-60 minutes. The topics are oral hygiene, medicine safe, living safe, food safe.
  Arms: Health education

SUMMARY:
Objective: The study aims to understand the physical function, body composition, mental state, behavior, depression, and life quality change of the elderly in a long-term care before and after the intervention. Four interventional activities are sitting strength training, games, sitting strength training with games, and health education.

DETAILED DESCRIPTION:
Expected results: (1) The program will facilitate arrange activities that are beneficial to the body and mind, activate bodily functions, and promote the quality of life of the elderly in Taiwan. (2) The program can compare the effectiveness of different trainings for the elderly and provide a reference for future implementation planning. (3) Evidence of the empirical study of this program can provide future comparisons with other domestic and foreign studies.

ELIGIBILITY:
1.Inclusion Criteria:

1. Elderly persons between the age of 60 and 100 who take long-term care of the relevant units do not have limited sports
2. stable condition with sufficient physical strength: at least one hour sitting in the wheelchair or bed edge.
3. Subjects in the past month tended to live in static state (less than 150 minutes of exercise time per week).

2.Exclusion Criteria:

1. Serious illness / unstable status (judged by medical staff), such as serious cardiopulmonary diseases, severe malignant tumor (assessment from medical personnel), severe malnutrition (mini nutrition assessment scale 0-7 points).
2. Unstable weight over the past six months (> ± 4 kg).

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2018-02-02 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
change from baseline body composition at 4 months and 8 months | baseline, 4 months, 8 months
  bioelectrical impedance analysis for body composition
change from baseline body function (ADL)at 4 months and 8 months | baseline, 4 months, 8 months
  The barthel index for activities of daily living
change from baseline muscle strength at 4 months and 8 months | baseline, 4 months, 8 months
  lb or kg
change from baseline quality of life at 4 months and 8 months | baseline, 4 months, 8 months
  WHOQOL-BREF scale for quality of life measurement from world health organization questionnaire.
change from baseline scale of quality of life at 4 months and 8 months | baseline, 4 months, 8 months
  EQ-5D (5 dimentions) scale for quality of life measurement from the EuroQol group.
change from baseline quality of life(dementia) at 4 months and 8 months | baseline, 4 months, 8 months
  QUALIDEM is a dementia-specific quality of life instrument.
change from baseline questionnaire of quality of life at 4 months and 8 months | baseline, 4 months, 8 months
  PERSONAL WELLBEING INDEX for quality of life measurement.
change from baseline body weight at 4 months and 8 months | baseline, 4 months, 8 months
  kg
change from baseline body height at 4 months and 8 months | baseline, 4 months, 8 months
  cm
change from baseline body function(IADL) at 4 months and 8 months | baseline, 4 months, 8 months
  Instrumental Activities of Daily Living for body function
change from baseline body function at 4 months and 8 months | baseline, 4 months, 8 months
  Body Awareness Rating Scale for body function

SECONDARY OUTCOMES:
change from baseline cognition at 4 months and 8 months | baseline, 4 months, 8 months
  The Clinical dementia rating scale (CDR) for memory, orientation, problem solving, community affairs, hobbies and personal care measurement.
change from baseline behavior at 4 months and 8 months | baseline, 4 months, 8 months
  The Cohen-Mansfield agitation inventory for aggressive behavior, physically nonaggressive behavior, verbally agitated behavior measurements.
change from baseline depression at 4 months and 8 months | baseline, 4 months, 8 months
  cornell scale for depression measurement: a score >10 probably major depressive episode ,A score >18 denote major depressive episode
change from baseline sleep(PSQI) at 4 months and 8 months | baseline, 4 months, 8 months
  The pittsburgh sleep quality index for sleep time and efficiency.
change from baseline mental and cognition at 4 months and 8 months | baseline, 4 months, 8 months
  Alzheimer's disease assessment scale(ADAS) for cognitive behavior, recall, recognition, constructional praxis measurement.
change from baseline mental at 4 months and 8 months | baseline, 4 months, 8 months
  Clock test for constructional measurement.
change from baseline sleep at 4 months and 8 months | baseline, 4 months, 8 months
  The actigraph for sleep time and efficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Ching Chiu, Phd, Study Chair — Instructor of Central Taiwan University of Science and Technology
Locations (1):
- Central Taiwan University of Science and Technology, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No